CLINICAL TRIAL: NCT05318716
Title: The Fat Analysis Trial (FAT): The Impact of Lip-aspirate Processing on Fat Resorption in Autologous Fat Grafting to the Breast: A Randomized Controlled Trial
Brief Title: The Fat Analysis Trial (FAT) - Assessing the Impact of Lipo-aspirate Processing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Tanya DeLyzer, Associate Professor, Division of Plastic and Reconstructive Surgery, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11811
Record Dates: First submitted 2022-03-24; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Breast Asymmetry; Fat Atrophy
Keywords: Fat grafting; Fat survival; Breast surgery
MeSH Terms: conditions — Anisomastia

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial, we aim to recruit patients already scheduled to undergo fat grafting to the breast for reconstruction or cosmetic augmentation.
Who Masked: Participant, Outcomes Assessor
Masking Description: When the patients check in at the reception desk, they will be assigned a ticket with a 0 or 1 sequentially. This will be placed in their file. Group 0 patients will receive Decantation, and group 1 will receive Revolve.
  The nurse will collect this ticket, along with the patient's registration documents to prepare the equipment.
  Photography will be done by a research assistant/coordinator. The person will be responsible for imaging patients, as well as conducting the volume analysis following training by the software manufacturer. This person will be blinded to which method is used.
  During subsequent follow ups, the patient will have a 0 or 1 in their chart, to accurately collect data while in follow up.
  The surgeon, assistants and nurses will not be able to be blinded as they are the person responsible for using the device in the operating room.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Reconstructive group (Experimental): This group of patients would be undergoing fat grafting following implant-based reconstruction. We will be excluding patients that have had autologous based reconstruction, including regional and free flaps. This group will be analyzed based on volume (<200cc or 50% and >200cc or 50%) as well as subgroup analysis based on adjuvant chemo or radiation therapy.
  Interventions: Device: Fat grafting - Revolve device; Device: Fat grafting - Decantation
- Cosmetic augmentation group (Experimental): This group of patients will be undergoing a primary or secondary augmentation for cosmesis. They will be included if this is a primary augmentation using fat grafting or a secondary augmentation with no history of fat grafting to the breasts.
  Interventions: Device: Fat grafting - Revolve device; Device: Fat grafting - Decantation

INTERVENTIONS:
Device: Fat grafting - Revolve device — Standardized fat collection The donor areas previously agreed on by the patient and surgeon for fat harvesting will be injected with pre-standardized formulae and volume of tumescent fluid, and fat will be extracted using a standardized harvesting method between surgeons. Once the fat is collected. It will then be processed in one of two ways depending on the patient's group, using a Revolve system or via decantation. Fat will then be injected into the breast using a 10 or 20cc syringe in the standard retrograde manner to achieve the desired size and shape. A standard gauze-based dressing will be applied post-operatively, with no compression.
Device: Fat grafting - Decantation — Standardized fat collection The donor areas previously agreed on by the patient and surgeon for fat harvesting will be injected with pre-standardized formulae and volume of tumescent fluid, and fat will be extracted using a standardized harvesting method between surgeons. Once the fat is collected. It will then be processed in one of two ways depending on the patient's group, using a Revolve system or via decantation. Fat will then be injected into the breast using a 10 or 20cc syringe in the standard retrograde manner to achieve the desired size and shape. A standard gauze-based dressing will be applied post-operatively, with no compression.

SUMMARY:
Fat grafting has been gaining popularity over the past decade. It is now commonly used for breast augmentation and reconstruction, however a major challenge remains the high rate and unpredictable rate of fat resorption post-operatively, leading to volume loss and patient dissatisfaction. Currently there is no consensus on the ideal technique to process donor fat to minimize the rate of resorption. Our study aims to compare two common processing methods to determine if one is superior for fat volume retention.

DETAILED DESCRIPTION:
Fat grafting is a technique used commonly in plastic surgery that has gained popularity in breast augmentation and breast reconstruction. This technique involves harvesting fat using liposuction from donor sites, processing the extracted fat and re-injecting it back into the breast for the desired volume and shape. Fat grafting has gained popularity due to its resulting natural appearance and feel. This technique can also be used in conjunction with implant reconstruction to achieve a more natural contour and symmetry. However, the main issue is a low rate of fat retention, which, based on the literature, is inconsistent and only an average of 60% of the volume of fat injected. Furthermore, there are very few clinical studies studying the long-term clinical survivability of the grafted fat. Therefore, care must be taken in setting patient expectations, and sometimes multiple sessions are required to achieve the desired results.

There are currently multiple techniques used in harvesting and processing fat for grafting, and it is unclear in the current literature if the processing technique used affects the level of fat resorption. General principles of fat grafting include gentle extraction to avoid damage and processing to remove excess infiltration fluid and impurities before injection. The fat is collected from donor areas for extraction, using either manual or power-assisted liposuction. For processing, several products and processing solutions have been developed in recent years, including the Revolve system (AbbVie/Allergan), which is currently used at our institution. Prior to these systems, simple decantation of fat by gravity or centrifugation was used. However, due to damage to fat during processing and lower retention rates in the literature, centrifugation has largely been abandoned as a processing method. However, there is no standard method of donor fat harvest or processing, and there is a lack of well-defined prospective clinical studies comparing popular techniques in the current literature, particularly in the long term. Additionally, the amount of fat injected and patient factors such as previous radiation can affect the amount of fat retention. Further in-vitro studies are required to clarify factors that affect fat survivability.

In order to assess the rate of fat retention in the breast, quantitative imaging tools have been validated in the literature. One of the most popular techniques is 3D body surface scans. These can be taken easily, quickly, and cost-effectively for volume assessment at various time points pre and postoperatively. Comparatively, MRI imaging is costly, time-consuming and therefore not practical for frequent follow-up. Furthermore, as 3D imaging becomes more accessible, its use could become more common in clinical practice for preoperative planning and objective assessment of outcomes.

Methods Aims Currently, there is a lack of prospective clinical studies directly comparing the rate of fat graft retention between processing techniques. Our primary outcome aims to compare two common processing methods; decantation and the Revolve system. Investigators will measure the retention rate using 3D imaging techniques (Vectra H2, Canfield), in the place of traditional 2D photography, for quantitative measurement of breast volume. Our secondary outcomes include the assessment of operating time, cost, and collect secondary outcomes related to surgical complications and outcomes. Investigators will tangentially perform a qualitative review of the patient's pre and post-operatively using the validated Breast-Q questionnaire. This study will be conducted at LHSC sites in London, Ontario.

ELIGIBILITY:
Inclusion Criteria:

* Any patient above the age of 18 undergoing fat grafting from any donor site to the breast for cosmetic or reconstructive purposes.
* We will accept patient who have an implant for either cosmetic or reconstructive purposes

Exclusion Criteria:

* Previous fat grafting
* Autologous breast reconstruction (regional or free flap)
* unable to consent to the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
1. What is the volume of fat retained between the two most common methods of fat processing? | 12 months recruitment and 24 months follow up
  Volume based Sub-division based on 3D volumetric analysis. Height (in metres) and weight (in kilograms) will be recorded to calculate BMI. This will be needed to assess weight stability during the follow up period.
  Each of the above groups will be stratified based on breast volume, as well as injected volume. Each group will be divided into low volume, which will be less than 200cc of injected fat or 50% of breast volume, whichever is greater. The high-volume group will include volumes greater than 200cc or 50% of breast volume.
  Imaging A Vectra H2 (Canfield medical, NJ) will capture a 3D image in place of our traditional 2D imaging, for both pre-operative and post-operative photos. A volumetric analysis will be performed using the proprietary software. With a pre-operative baseline volume, we will be able to track fat survival between the two-methods post-operatively during follow up visits.
  Total follow up time will be 24 months post-operatively.
How satisfied are the patients between each method of fat grafting? | 36 months total
  We will tangentially perform a qualitative review of the patient's pre and post-operatively using the validated Breast-Q questionnaire. The BREAST-Q module for women who undergo breast augmentation is a rigorously developed PROM that is comprised of 9 independently functioning scales. It has undergone extensive psychometric evaluation and its developers report that it may be used like interval-scale data. Scores from these instruments are scaled to range from 0 to 100. This study will be conducted at affiliated clinical sites in London, Ontario.

SECONDARY OUTCOMES:
3. Does one method of fat processing have a reduced rate of short, or long term complications? | 36 months
  the assessment of operating time (recorded in minutes) from the time tumescence is injected, until the injecting is complete. The additional cost of the device will be accounted for in the analysis (in US dollars), and collect secondary outcomes related to surgical complications and outcomes. These will be recorded prospectively and classified into minor and major, where major would be considered if needing surgery to correct an issue.

OTHER OUTCOMES:
Is the grafted fat incorporated better between the two methods? | 3 months
  We will include a bedside ultrasound (US) image of the breast tissue at 3 months, to assess fat incorporation and the amount of oil and oil cysts. US images will be taken bedside, with a visual analysis of the images done by a blinded assessor.
  It will be measured with a visual analog scale from 0 to 5, with 0 representing no oil cysts and 5 representing an abundance of oil cysts. The assessors will be two different blinded plastic surgeons.

IPD SHARING:
Plan to Share IPD: Undecided
This is an ongoing discussion. At present there is a slight lean towards not making individual participant data available. This is to protect patient information during inclusion in this trial.